CLINICAL TRIAL: NCT01485952
Title: An Exploratory Clinical Trial in Early Stage Huntington's Disease Patients to Assess Pharmacokinetics, Candidate Pharmacodynamic Measures of Target Engagement and Disease Modulation as Well as Acute Phenotypical Effects Following Multiple Oral Doses of SEN0014196.
Brief Title: An Exploratory Clinical Trial in Early Stage Huntington's Disease Patients With SEN0014196
Acronym: PADDINGTON
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Siena Biotech S.p.A. (Industry)
Collaborators: Seventh Framework Programme (Other); European Huntington's Disease Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S015-004; CTA Number: 2010-021563-32 (Other Grant/Funding Number: European Commission 7th Framework Programme)
Record Dates: First submitted 2011-11-29; First posted 2011-12-06 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Huntington Disease
Keywords: Huntington Disease; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Dementia; Chorea; Dyskinesias; Movement Disorders; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Genetic Diseases, Inborn; Cognition Disorders; Mental Disorders
MeSH Terms: conditions — Huntington Disease; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Dementia; Chorea; Dyskinesias; Movement Disorders; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Genetic Diseases, Inborn; Cognition Disorders; Mental Disorders | interventions — 6-chloro-2,3,4,9-tetrahydro-1H-carbazole-1-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SEN0014196 (Low Dose) (Experimental): 10 mg, once daily administration (immediate release capsule)
  Interventions: Drug: SEN0014196 (Low Dose)
- SEN0014196 (High dose) (Experimental): 100 mg, once daily administration (immediate release capsule)
  Interventions: Drug: SEN0014196 (High Dose)
- Placebo (Placebo Comparator): Once daily (immediate release capsule)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEN0014196 (Low Dose) — 10 mg once daily administration (immediate release capsule)
  Arms: SEN0014196 (Low Dose)
Drug: SEN0014196 (High Dose) — 100 mg once daily administration (immediate release capsule)
  Arms: SEN0014196 (High dose)
Drug: Placebo — Once daily administration (immediate release capsule)
  Arms: Placebo

SUMMARY:
The primary objective of this study is to provide biological samples from patients with Huntington's disease to allow characterisation of the pharmacological mechanism of action of SEN0014196.

DETAILED DESCRIPTION:
This study will establish the acute phenotypical and biological effects of repeated dose application of SEN0014196 in patients with Huntington's disease, providing biomaterials for biomarker studies (levels of circulating huntingtin, acetylation status of mutant huntingtin, innate immune markers, transcriptional profiles). Evaluation of phenotypic effects will include UHDRS scores, total functional capacity. Safety assessments will include ECG, vital signs, laboratory safety tests and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early Huntington's Disease (age: 18 to 70 years), i.e. genetically confirmed (CAG repeat length ≥36) HD, motor signs of HD (motor score of the UHDRS > 5) and a TFC of ≥7.
* All patients will have a body weight greater than 50 kg.
* Female subjects must be surgically sterile or post-menopausal, no spontaneous menstruation for at least one year before the first dose, non-lactating and have a negative urine pregnancy test. Male subjects participating in the trial and their female contraception from the time of taking the first dose of the study drug until three months after taking the last dose. This must include a condom or other barrier method.
* All subjects must be capable of providing written informed consent.
* Subjects must have no clinically significant and relevant history that could affect the conduct of the study and evaluation of the data, as ascertained by the Investigator through detailed medical history and screening assessments.

Exclusion Criteria:

* Participation in a study of an investigational drug within 30 days of the baseline visit.
* Subjects with presence of psychosis and/or confusional states.
* Subjects with clinically significant laboratory or ECG abnormalities at Screening.
* Subjects with clinically relevant hematological, hepatic, cardiac or renal disease.
* A medical history of infection with human immunodeficiency virus, hepatitis C and/or hepatitis B.
* Any relevant condition, behaviour, laboratory value or concomitant medication which, in the opinion of the Investigator, makes the subject unsuitable for entry into the study.
* Subjects who have previously received histone deacetylase inhibitors e.g. vorinostat or have participated in a clinical trial using compound suspected of interfering with protein acetylation status.
* A history of malignancy of any type within 2 years prior to screening. A history of surgically excised nonmelanoma skin cancers is permitted.
* Subjects with a significant history of drug allergy as determined by the Investigator.
* Subjects who have a significant history of alcoholism or drug/chemical abuse as determined by the Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the change from baseline of a series of pharmacodynamic markers in peripheral blood mononuclear cells | Baseline, Day 7, Day 14, Follow-Up
  Collection of peripheral blood mononuclear cells for biomarker investigations, specifically acetylation status of mutant huntingtin, levels of circulating huntingtin, innate immune markers and transcriptional profiles

SECONDARY OUTCOMES:
To determine the safety and tolerability following repeated doses of SEN0014196 over two weeks at two dose levels in patients with Huntington's disease | Baseline, Day 7, Day 14, Follow-up
  Safety assessments will include ECG, vital signs, laboratory safety tests, and physical and neurological examination. Tolerability will include type and frequency of adverse events.
To determine the pharmacokinetics of repeated doses of SEN0014196 at two dose levels when administered over two weeks in patients with Huntington's disease | Baseline, Day 14
  The following parameters will be assessed: maximum observed plasma concentration (Cmax), time of maximum observed plasma concentration(tmax), AUC from time zero to the length of the dosing interval (tau) (AUC0-τ), AUC from time zero to the last quantifiable concentration (AUC0-last), AUC from time zero to infinity (AUC0-∞), terminal elimination half-life (t1/2), and terminal elimination rate constant (λz). Gender differences. Dose proportionality.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard G Landwehrmeyer, MD, PhD, Principal Investigator — European Huntington's Disease Network
Locations (1):
- Universitätsklinik Ulm, Neurologie, Ulm, Germany